CLINICAL TRIAL: NCT01952561
Title: An Open-label, Parallel-group Pharmacokinetic Trial in Healthy HIV-negative Women to Characterize the Release Profile of Dapivirine Delivered by a Silicone Matrix Ring (Ring 004), Containing 25 mg of Dapivirine, Over Various Ring Use Periods
Brief Title: Expanded Use PK of Dapivirine Vaginal Ring
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: International Partnership for Microbicides, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IPM 034
Record Dates: First submitted 2013-09-17; First posted 2013-09-30 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2013-09

CONDITIONS: Pharmacokinetics
Keywords: pharmacokinetics; vaginal ring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- 2 weeks (Experimental)
  Interventions: Drug: dapivirine ring
- 1 week (Experimental)
  Interventions: Drug: dapivirine ring
- 4 weeks (Experimental)
  Interventions: Drug: dapivirine ring
- 8 weeks (Experimental)
  Interventions: Drug: dapivirine ring
- 12 weeks (Experimental)
  Interventions: Drug: dapivirine ring

INTERVENTIONS:
Drug: dapivirine ring

SUMMARY:
Study will evaluate the vaginal and blood pharmacokinetics of dapivirine from a vaginal ring containing 25 mg worn for 1, 2, 4, 8 or 12 months.

ELIGIBILITY:
Key Inclusion Criteria:

1. Women 18 and ≤ 40 years of age who can give written informed consent
2. Available for all visits and consent to follow all procedures scheduled for the trial
3. Healthy, based on medical history, vital signs, physical examination, urinalysis, laboratory evaluations for genital infections, and laboratory evaluations for haematology and chemistry
4. HIV-negative as determined by an HIV test at the time of enrolment
5. On a stable form of contraception, defined as:

   * A stable oral contraceptive regimen for at least 2 months prior to enrolment, OR
   * Transdermal contraceptive patch for at least 3 months prior to enrolment, OR
   * Long-acting progestins for at least 6 months prior to enrolment, OR
   * An IUD inserted at least 3 months prior to enrolment, OR
   * Have undergone surgical sterilisation at least 3 months prior to enrolment AND willing to use oral contraceptives if necessary to delay menstruation during the vaginal sampling period
6. Upon pelvic examination at the time of enrolment, the cervix and vagina appear normal as determined by the Investigator/Physician
7. Asymptomatic for genital infections at the time of enrolment
8. Willing to refrain from the use of topical vaginal medications, vaginal products or objects
9. Documentation of no abnormality on cervical cytology, including grossly bloody smear, within 90 days prior to screening
10. Willing to refrain from participation in any other research trial for the duration of this trial
11. Willing to provide adequate locator information for trial retention purposes and be reachable per local standard procedures, e.g. by home visit or telephone, or via family or close neighbour contacts
12. Willing to agree to abstain from all the following for a total of 2 days (48 hours) prior to each trial visit:

    * Penile-vaginal intercourse
    * Oral contact with her genitalia
13. Hepatitis B and C negative at the time of enrolment.

Key Exclusion Criteria:

1. Currently pregnant or had their last pregnancy outcome within 3 months prior to screening
2. Currently breast-feeding
3. Currently or within two months of participation in any other clinical research trial involving investigational or marketed products prior to screening
4. Untreated symptomatic urogenital infections, e.g. urinary tract or other sexually transmitted infections, or other gynaecological conditions such as vaginal itching, pain, or discharge, within 2 weeks prior to enrolment
5. Have a Grade 2 or higher pelvic examination finding, according to the DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events;
6. History of significant urogenital or uterine prolapse, undiagnosed vaginal bleeding, urethral obstruction, incontinence or urge incontinence
7. Current vulvar or vaginal symptoms/abnormalities that could influence the trial results
8. Cervical cytology at screening that requires cryotherapy, biopsy, treatment (other than for infection), or further evaluation
9. Symptomatic genital herpes simplex virus (HSV) infection or a history of genital herpetic infection
10. Any Grade 2, 3 or 4 haematology, biochemistry or urinalysis laboratory abnormality at baseline (screening) according to the DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events;
11. Unexplained, abnormal bleeding per vagina during or following vaginal intercourse, or gynaecologic surgery within 90 days prior to enrolment
12. Any history of anaphylaxis or severe allergy resulting in angioedema; or a history of sensitivity/allergy to latex or silicone
13. Any serious acute, chronic or progressive or signs of cardiac disease, renal failure, or severe malnutrition
14. Have undergone a hysterectomy
15. Any condition(s) that, in the opinion of the Investigator, might interfere with adherence to trial requirements or evaluation of the trial objectives.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2013-11; Primary Completion 2014-03 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
dapivirine pharmacokinetics in plasma | 1,2,4,8 or 12 weeks